CLINICAL TRIAL: NCT04760496
Title: Effect of Increased Oxytocin Doses on the Mode of Delivery in Obese Primiparous Women With Spontaneous or Induced Labour. A Double-blind, Randomised, Controlled Trial
Brief Title: Effect of Increased Oxytocin Doses on the Mode of Delivery in Obese Primiparous Women With Spontaneous or Induced Labour
Acronym: PROXYMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-002640-23
Record Dates: First submitted 2021-01-29; First posted 2021-02-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-08

CONDITIONS: Obese; Primiparous Women; Oxytocin
Keywords: Obese; Primiparous women; Oxytocin
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: There is two group of patient for which the prescription of oxytocin is required for the care :
  the control group will receive will receive oxytocin at 2 mIU/mL (standard dose) the experimental group will receive oxytocin at 4 mIU/mL
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An "out-of-protocol" healthcare professional (midwife / nurse) will prepare oxytocin. The "out-of-protocol" healthcare professional (midwife / nurse) will not be a study's investigator, and will not be involved in the patient's care. The randomization group will not be communicated to the investigator or any medical personnel involved in the study or patient by the "out-of-protocol" nurse/midwife, in order to preserve the double-blind design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive oxytocin at 4 mIU/mL
  Interventions: Drug: Oxytocin 4 mIU/mL
- Control group (Active Comparator): The control group will receive oxytocin at 2 mIU/mL
  Interventions: Drug: Oxytocin 2 mIU/mL

INTERVENTIONS:
Drug: Oxytocin 4 mIU/mL — Oxytocin at 4 mIU/mL administrated by IV infusion controlled by pump or electric syringe.
  Arms: Experimental group
Drug: Oxytocin 2 mIU/mL — Oxytocin at 2 mIU/mL administrated by IV infusion controlled by pump or electric syringe.
  Arms: Control group

SUMMARY:
The rate of caesarean section is higher among obese pregnant women, leading to increased morbidity in this already vulnerable population. Oxytocin is the main drug used in obstetrics to optimize progress of labour, but observational studies have suggested that its efficiency may be insufficient in obese women with usual doses.

We design a randomised controlled trial to test the effect of an increased oxytocin dose on the rate of caesarean section in obese primiparous women with spontaneous or induced labour.

DETAILED DESCRIPTION:
The hypothesis underlying this trial is that an increase in oxytocin dose can reduce the rate of caesarean sections in primiparous obese patients, with a spontaneous or induced onset of labour, without increasing maternal or neonatal morbidity. This would be a major step forward in reducing morbidity in an at-risk population and in improving the obstetric prognosis for future pregnancies.

The research is a double-blind controlled trial, including primiparous obese women in spontaneous or induced labour, for whom a prescription of oxytocin is decided. Oxytocin is currently indicated for notably "insufficiency of uterine contractions, at the beginning or during labour".The recommended dosage in the market authorization will be used for the control group.

The control group will receive oxytocin at 2 milli-International unit /mL and the intervention group at 4 milli-International unit /mL, controlled by pump (final volume = 500 mL) or electrical syringe (final volume = 50 mL).

The primary objective is to compare the effect of higher doses of oxytocin (intervention group) vs standard doses of oxytocin (control group) on the rate of caesarean sections in obese patients with spontaneous or induced onset of labour.

The secondary objectives will be to compare the effect of higher doses of oxytocin (intervention group) vs standard doses of oxytocin (control group) on maternal and labour complications (length of labour, arrest of labour, interruption of oxytocin perfusion and reason, uterine hyper-stimulation, mode of vaginal delivery, reason for caesarean section, post-partum haemorrhage, maternal blood transfusion, volume of oxytocin infusion, oxytocin side effects), as well as foetal complications and neonatal complications.

ELIGIBILITY:
Inclusion criteria

Inclusion criteria are the following:

* Age ≥ 18 years
* Nulliparous (no previous childbirth beyond 22 SA)
* BMI ≥ 30 kg/m² at the beginning of pregnancy
* Singleton pregnancy
* Spontaneous or induced onset of labour
* Cephalic presentation
* Term ≥ 37 weeks of gestation and < 42 weeks of gestation
* Medical Indication and absence of medical contraindication for oxytocin during labour: inadequate and/or ineffective uterine contraction and/or delayed cervical dilation
* Written consent
* Affiliation to a french social security system

Exclusion criteria

Exclusion criteria are the following:

* Hypersensitivity to the active substance (oxytocin), to any of its excipients or to latex (risk of cross allergy)
* Medical contraindication for oxytocin
* Coagulation disorders
* Foetal growth restriction (inferior to 5th percentile)
* Foetal malformation (major)
* Foetal heart rate anomalies before use of oxytocin (at the time of inclusion)
* History of uterine surgery (scarred uterus of gynaecological origin)
* Patient with a disease requiring caesarean section prior to labour (planned caesarean section before labour)
* Severe renal failure
* Patient deprived of their liberty (under curatorship or guardianship)
* Participation in another interventional trial of category 1. Patients included in interventional research with minimal risk and constraints may participate in the study after the investigator's assessment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 443 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of caesarean section during labour | through study completion, an average of 1 month
  The decision of caesarean section is made by the responsible obstetrician in charge of the patient, he or she will be blinded of the patient's group (oxytocin dosage) to avoid differential indication for caesarean section.
  Therefore, the decision to perform (or not) a caesarean section will be only based on foetal/maternal criteria, independently of oxytocin dosage.

SECONDARY OUTCOMES:
Length of labour phases | Through study completion, an average of 1 month
  Length of labour phases is measured in minutes (from 2 cm of dilation until delivery)
Arrest of labour | Through study completion, an average of 1 month
  It will be evaluated if there is two or more hours without cervical dilation (yes/no)
Interruption of oxytocin perfusion and causes | through study completion, an average of 1 month
  Interruption of oxytocin perfusion (yes/no) and causes (foetal heart anomalies / uterine hyperkinesia / uterine hypertonia / other)
Uterine hyper-stimulation | Through study completion, an average of 1 month
  Uterine hyper-stimulation (more than 5 uterine contractions per 10 min)
Mode of vaginal delivery | Through study completion, an average of 1 month
  Spontaneous or operative delivery.If operative vaginal delivery: indication
Reason for the caesarean section | through study completion, an average of 1 month
  foetal heart anomalies / labour arrest / other
Post-partum haemorrhage | Through study completion, an average of 1 month
  Post-partum haemorrhage (yes/no) and its volume (mL). Post-partum haemorrhage is defined as blood lost ≥ 500 mL in the 2 hours after birth.
Maternal blood transfusion | Through study completion, an average of 1 month
  Maternal blood transfusion (yes/no) (for the duration of the hospitalization)
Volume of oxytocin infusion | Through study completion, an average of 1 month
  Volume of oxytocin infusion (mL/H)
Oxytocin side effects | Through study completion, an average of 1 month
  nausea, vomiting, headaches, increased or decreased heart rate, allergic reaction, skin rash
Foetal complications | Through study completion, an average of 1 month
  * Foetal heart rate anomalies requiring second-line monitoring (as pH/lactate blood test at scalp) or emergency delivery (yes / no)
  * Appearance of meconium (yes / no)
  * Chorioamnionitis (yes/no): defined as the combination of 2 of the next 3 signs: maternal fever more than 38°5 during labour and/or foetal heart tachycardia and/or biological infection sign
Neonatal complications | Through study completion, an average of 1 month
  * Apgar score at 5 min
  * Umbilical arterial cord pH
  * Neonatal resuscitation (yes / no): defined by at least artificial ventilation
  * Transfer to neonatal care unit (yes / no)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra BENACHI, PHD, MD, Principal Investigator — Antoine Béclère Hospital, APHP
Locations (12):
- France (12):
  - CHU d'Angers, Angers
  - CHU de Bordeaux (Pellegrin), Bordeaux
  - Hôpital Béclère, Clamart
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU de Montpellier, Montpellier
  - CHU de Nimes, Nîmes
  - Hôpital Cochin Port Royal, Paris
  - Hôpital Tenon, Paris
  - CHU de Poissy St Germain, Poissy
  - CHU de Saint Etienne, Saint-Etienne
  - CHU de Strasbourg (Centre Médico Chirurgical et Obstétrical), Schiltigheim
  - CHU de Strasbourg (Hôpital de Hautepierre), Strasbourg